CLINICAL TRIAL: NCT06679582
Title: A Phase 1/2, Open-label Study Evaluating the Efficacy, Safety, and Pharmacokinetics (PK) of Luveltamab Tazevibulin (STRO-002) in Infants and Children < 12 Years of Age With CBFA2T3::GLIS2 Acute Myeloid Leukemia (AML)
Brief Title: Luveltamab Tazevibulin (STRO-002) in Infants and Children < 12 Years of Age With Relapsed/Refractory CBFA2T3::GLIS2 AML
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Terminated Early
Sponsor: Sutro Biopharma, Inc. (Industry)
Collaborators: Children's Oncology Group (Network); Innovative Therapies For Children with Cancer Consortium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REFRαME P1; 2023-506240-16-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-02; First posted 2024-11-07 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2024-11

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: CBFA2T3::GLIS2 Fusion; CBFA2T3::GLIS2 AML; RAM Phenotype (CD56pos); CD45, CD38, HLA-DR weak or absent); REFRaME; AML, Child; Pediatric AML; REFRaME-P1; Luveltamab; tazevibulin; STRO-002
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: This trial has two parts, Part 1 will use a parallel model by assessing two luveltamab tazevibulin doses (3.5 and 4.3 mg/kg every 2 weeks). Two cohorts will be run in parallel. The transition from part 1 to part 2 is sequential, with part 2 testing the dose selected at the end of part 1.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort 1 (Experimental): Luveltamab tazevibulin 3.5mg every 2 weeks
  Interventions: Drug: Luveltamab tazevibulin
- Cohort 2 (Experimental): Luveltamab tazevibulin 4.3 mg every 2 weeks
  Interventions: Drug: Luveltamab tazevibulin

INTERVENTIONS:
Drug: Luveltamab tazevibulin — Luveltamab tazevibulin is an antibody-drug conjugate (ADC) targeting folate receptor α (FRα or FOLR1). It consists of an IgG1 antibody (SP8166) conjugated to cathepsin cleavable 3-aminophenyl hemiasterlin payload, yielding a homogenous ADC with a drug antibody ratio of four. The active warhead (SC209) inhibits tubulin polymerization leading to mitotic arrest and cell death.
  Other Names:
  * STRO-002
  * Luvelta
  Other Names: STRO-002; Luvelta

SUMMARY:
This trial will evaluate whether luveltamab tazevibulin is well tolerated and active against a rare form of AML carrying a particular genetic abnormality called CBFA2T3::GLIS2 that arises in infants and children. To be treated in this trial children must have a leukemia which did not respond or recurred after prior treatment. Luveltamab tazevibulin is an antibody-drug conjugate, which brings tazevibulin, an anticancer drug, to a molecule called FOLR1, present on the surface of CBFA2T3::GLIS2 AML cells.

DETAILED DESCRIPTION:
This is a registrational international, multicenter, two-part open label Phase 1/2 trial in an extremely rare pediatric disease (around 17 new patients a year in US and 10 in EU). Part 1 randomizes subjects 1:1 to one of two luveltamab tazevibulin dose cohorts (1a and 1b). Part 2 further evaluates the safety and the efficacy of the selected dose. Subjects who achieve complete remission after two cycles of treatment may continue luveltamab tazevibulin as monotherapy, while non-responders at PI discretion may add luveltamab tazevibulin with standard of care (SOC) AML treatments. Luveltamab tazevibulin is given IV every two week as monotherapy and every 4 weeks when given with chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* AML with CBFA2T3::GLIS2 gene fusion centrally confirmed
* Refractory or relapsed disease with ≥ 5% bone marrow involvement with leukemic blasts by morphology
* Age < 12 years.
* Lansky performance of ≥ 50
* Adequate organ functions

Exclusion Criteria:

* Active central nervous system (CNS) disease (CNS3)
* Pre-existing clinically significant corneal disorders or constitutional diseases associated with an increased risk of AML treatment toxicities
* Active or uncontrolled infections or other active severe intercurrent illnesses,
* Prior treatment with a FOLR1- targeting ADCs or with ADCs that contain a tubulin inhibitor
* History of allogeneic hematopoietic stem cell transplant or any organ transplant in the prior 84 days
* Graft versus host disease (GVHD) of any grade or GVHD treatment with exception of low dose steroids

Ages: 1 Day to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2024-12-04 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Evaluate efficacy of luveltamab tazevibulin monotherapy | Up to 12 weeks
  Complete remission rate

SECONDARY OUTCOMES:
Assess additional efficacy outcome measures | Up to 2 years
  • Duration of CR
Evaluate safety measures | Up to 2 years
  Incidence and severity of AEs and clinical laboratory abnormalities per NCI CTCAE v5.0 in patients receiving luveltamab tazevibulin monotherapy.
To characterize the PK of luveltamab tazevibulin | Up to 2 years
  Concentration of luveltamab tazevibulin (ADC, TAb, and SC209) in the blood.
Assess the immunogenic potential of luveltamab tazevibulin | Up to 2 years
  Incidence of ADAs
Assess additional efficacy outcome measures | Up to 2 years
  • Response rate including complete remission with partial hematologic recovery (CRh) rate [CR = CRh]
Assess additional efficacy outcome measures | Up to 2 years
  • Event-free survival (EFS)
Assess additional efficacy outcome measures | Up to 2 years
  • Relapse-free survival (RFS)
Assess additional efficacy outcome measures | Up to 2 years
  • Overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Berman, MD, Study Director — Sutro Biopharma
Locations (36):
- United States (23):
  - Childrens Hospital of Alabama, Birmingham, Alabama
  - Childrens Hospital of Los Angeles, Los Angeles, California
  - Lucile Packard Childrens Hospital-Stanford, Palo Alto, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - Childrens National Hospital, Washington D.C., District of Columbia
  - Children's Hospital of Atlanta-Emory, Atlanta, Georgia
  - Ann & Robert H. Lurie Childrens Hospital, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Minnesota-Masonic Cancer Center, Minneapolis, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Washington University-School of Medicine, St Louis, Missouri
  - Columbia University Irving Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine-Dan Duncan Comprehensive Cancer Center, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Massey Cancer Center-Adult Outpatient Pavillion, Richmond, Virginia
  - Seattle Childrens, Seattle, Washington
- St Anna Kinderspital, Vienna, Austria
- Canada (2):
  - The Hospital for Sick Children, Toronto, Ontario
  - Centre Hospitalier Universitaire-Sainte Justice, Montreal, Quebec
- Rigshopitalet-University of Copenhagen, Copenhagen, Denmark
- France (2):
  - Institut d'hématologie et d'oncologie pédiatrique, Lyon
  - Hopital Armand Trousseau, Paris
- Germany (2):
  - Charite-Universitatsmedizin Berlin, Berlin
  - Universitatsklinikum-Essen, Essen
- Italy (2):
  - Fondazione IRCCS San Gerardo dei Tintori, Monza
  - Children Hospital Bambino Gesu IRCCS, Rome
- Princess Maxima Center for Pediatric Oncology, CS Utrecht, Netherlands
- Spain (2):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Infantil Universitario Nino Jesus-Servicio de Hematologia, Madrid

IPD SHARING:
Plan to Share IPD: No